CLINICAL TRIAL: NCT07400094
Title: Prospective Non-Randomized Phase II Study of Neoadjuvant Camrelizumab Combined With Paclitaxel and Carboplatin in Patients With Resectable Locally Advanced Squamous Cell Carcinoma of the Oral Cavity and Larynx (Stage III-IVA)
Brief Title: Neoadjuvant Chemoimmunotherapy (Camrelizumab + Paclitaxel + Carboplatin) for Resectable HNSCC
Acronym: NeoCamre-HN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Medical Research Radiological Centre of the Ministry of Health of Russia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoCamre-HN-01; LEC #1187/132 (Other: Local Ethics Committee, P.A. Hertsen)
Record Dates: First submitted 2026-01-29; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Laryngeal Neoplasms; Oral Cavity Neoplasm
Keywords: Head and Neck Squamous Cell Carcinoma; Neoadjuvant Therapy; Camrelizumab; Paclitaxel; Carboplatin; Pathological Complete Response; PD-1 Inhibitor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Laryngeal Neoplasms; Mouth Neoplasms | interventions — camrelizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Chemoimmunotherapy (Experimental): Patients receive 3 cycles of camrelizumab + paclitaxel + carboplatin followed by surgery.
  Number of Participants: 50 (Anticipated)
  Interventions: Drug: Camrelizumab; Drug: Paclitaxel; Drug: carboplatin; Procedure: Radical Surgery

INTERVENTIONS:
Drug: Camrelizumab — 200 mg IV on Day 1, every 21 days for 3 cycles
  Other Names: SHR-1210
Drug: Paclitaxel — 175 mg/m² IV on Day 1, every 21 days for 3 cycles
  Other Names: Taxol
Drug: carboplatin — AUC 6 IV on Day 1, every 21 days for 3 cycles
  Other Names: Paraplatin
Procedure: Radical Surgery — Standard radical resection 4-6 weeks after neoadjuvant therapy

SUMMARY:
This phase II study evaluates the efficacy and safety of neoadjuvant chemoimmunotherapy consisting of camrelizumab (PD-1 inhibitor), paclitaxel, and carboplatin in patients with resectable locally advanced (Stage III-IVA) squamous cell carcinoma of the oral cavity and/or larynx.

Fifty patients will receive 3 cycles of therapy (camrelizumab 200 mg IV, paclitaxel 175 mg/m2 IV, carboplatin AUC6 IV, Day 1 every 21 days) followed by radical surgery 4-6 weeks later. Patients are then stratified to risk-adapted adjuvant therapy based on pathological findings (radiation or chemoradiation with cisplatin if adverse features present).

The primary endpoint is the pathological complete response (pCR) rate and major pathological response (MPR, <10% viable tumor cells) rate at surgery. Secondary endpoints include objective response rate (ORR) by imaging (MRI/PET-CT), correlation of PET-CT metabolic response with pathological response, proportion requiring adjuvant chemoradiation, and 3-year event-free survival compared to historical controls.

Study period: 2026-2029.

DETAILED DESCRIPTION:
Investigator-initiated, single-arm, phase II study conducted at P.A. Hertsen Moscow Oncology Research Institute. Protocol approved by Local Ethics Committee (#1187/132).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the oral cavity and/or larynx, Stage III-IVA (cT1-2N1-2M0, cT3-4aN0-2M0)
* Resectable disease planned for surgical treatment
* Age 18-75 years
* No prior antitumor therapy for the current diagnosis
* Tumor sample available for PD-L1 expression assessment
* No other malignancies in anamnesis (except basal cell carcinoma of skin and carcinoma in situ of cervix)
* Absence of comorbidities preventing systemic chemotherapy and immunotherapy

Exclusion Criteria:

* Patient refusal to undergo planned treatment
* Protocol violations not related to medical indications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate | At the time of surgery (approximately 10-12 weeks from baseline)
  Rate of complete pathological response (absence of viable tumor cells in resected specimen)
Major Pathological Response (MPR) Rate | At the time of surgery (approximately 10-12 weeks from baseline)
  Rate of major pathological response (<10% viable tumor cells in resected specimen)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | After 3 cycles of neoadjuvant therapy (approximately 9 weeks)
  Rate of objective response by imaging (MRI/PET-CT) compared to historical TPF control
3-Year Event-Free Survival (EFS) | 3 years from enrollment
  EFS compared to historical control (surgery + RT/CRT)
Incidence of Adverse Events | From first dose until 30 days after surgery
  Safety profile compared to standard TPF induction chemotherapy
Proportion Requiring Adjuvant Chemoradiation | At the time of surgery
  Patients needing post-op CRT due to adverse pathological features vs historical control

CONTACTS AND LOCATIONS:
Overall Officials: Larisa V. Bolotina, MD, PhD, Study Chair — P.A. Hertsen Moscow Oncology Research Institute
Locations (1):
- P.A. Hertsen Moscow Oncology Research Institute, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
This is an investigator-initiated, single-center study conducted in Russia. Individual participant data will not be shared due to patient confidentiality requirements and institutional data protection policies.

REFERENCES:
- [Background] Wu D, Li Y, Xu P, Fang Q, Cao F, Lin H, Li Y, Su Y, Lu L, Chen L, Li Y, Zhao Z, Hong X, Li G, Tian Y, Sun J, Yan H, Fan Y, Zhang X, Li Z, Liu X. Neoadjuvant chemo-immunotherapy with camrelizumab plus nab-paclitaxel and cisplatin in resectable locally advanced squamous cell carcinoma of the head and neck: a pilot phase II trial. Nat Commun. 2024 Mar 11;15(1):2177. doi: 10.1038/s41467-024-46444-z. PMID 38467604